CLINICAL TRIAL: NCT05587595
Title: Transition From Paediatric Intensive Care to General Paediatrics and Pneumology Units : a Study of the Post-intensive Care Syndrome
Acronym: Presage-SPSI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP220341; IDRCB: 2022-A00267-36 (Registry Identifier: Ministry of health)
Record Dates: First submitted 2022-10-17; First posted 2022-10-20 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2022-10

CONDITIONS: Pediatric Post-intensive Care Syndrome; Intensive Care Unit Syndrome
Keywords: critical care; PICS
MeSH Terms: interventions — Surveys and Questionnaires; Data Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- children with complicated sickle cell disease hospitalised in pediatric intensive care unit (PICU)
  Interventions: Other: questionnaires & data collection
- children with complicated sickle cell disease hospitalised but not in intensive care unit
  Interventions: Other: questionnaires & data collection

INTERVENTIONS:
Other: questionnaires & data collection — questionnaires
  Other Names: questionnaires

SUMMARY:
In developed countries, mortality rates in pediatric intensive care units (PICUs) are around 4% and most children admitted to these units survive. However, some pediatric survivors experience long-term morbidity (cognitive, psychological and/or physical impairment) associated with their PICU stay and there is increasing awareness of the onset of post-intensive care syndromes (PICS) like in adults. However comprehensive descriptive data are still lacking regarding PICS in pediatrics (PICS-p).

The aim of this study is to describe (in nature and frequency) the alterations in health defined by the WHO of children who have passed through the PICU and constitute a possible PICS-p.

In order to do this, we will perform a prospective cohort study in Robert-Debré University Hospital including the PICU. We will include children with an unplanned hospitalization for more than 72 hours for acute complication of sickle cell disease (such as acute chest syndrome or vaso-occlusive crisis), acute asthma or sepsis and aged from 3 to 17 years. We plan to include 40 patients admitted to the PICU as well as 40 controls admitted to the general pediatrics unit or the pneumology unit without PICU admission, matched on diagnosis, age range and period.

The primary endpoint will be the prevalence of children that had been admitted to PICU and reporting cognitive, psychological, physical and social impairments measured by questionnaire and medical record data collection on the day before discharge and at the routine post-hospitalization visit.

Secondary objectives will be to study the risk factors for PICS-p, to compare alterations in cognitive, psychological, physical and social domains in children with the same diagnosis and age not admitted to the PICU during their hospitalization.

In order to this, we will measure the association with the PICU stay characteristics, parental experience and social characteristics of families. We will also report the prevalence of children not admitted in intensive care and reporting cognitive, psychological, physical and social impairments measured by questionnaire and medical record data collection on the day before discharge and at the routine post-hospitalization visit.

Patients and their parents will be given questionnaires the day before discharge and during the first follow-up consultation between 2 and 4 months after hospital discharge.

Questionnaires will include the Pediatric Symptom Checklist long version (Assessment of cognitive, psychological and social domains - 35 items scored from 0 to 2) reported by parents for children under 8 years and by the patients for children older than 8 years. older), the physical items of Pediatric Quality of Life scale (8 items scored from 0 to 4) and a parent self-questionnaire (including relationship to child, annual income, household composition, understanding and use of the French language, highest diploma of mother and father, social support (""How many people can you really count on when you need help?"")) and a parental mental health self-assessment (PHQ-8).

The analyses will be descriptive (description of the nature and frequency of alterations) and comparative (between children who have or have not been in PICU). Univariate tests will be performed to identify possible risk factors for post intensive care syndrome. Statistics will be carried out on SAS 9.4 software.

DETAILED DESCRIPTION:
Several large databases report mortality rates around 4% in pediatric intensive care units (PICUs) in developed countries, indicating that most children admitted to these units survive. Some pediatric survivors experience long-term morbidity associated with their PICU care, but comprehensive descriptive data are lacking.

In 2010, the Society of Critical Care Medicine (USA) organized a working group to raise awareness of long-term cognitive, psychological and physical impairments in adult ICU survivors. Impairments in these three domains are collectively referred to as Post-Intensive Care Syndrome ""PICS"". In the adult population, PICS affects 50-70% of ICU survivors, and its effects may persist for 5-15 years after ICU hospitalization. In adults, recovery and quality of life after ICU stay has been described by the World Health Organization.

In pediatrics, the framework of the pediatric post-intensive care syndrome ""PICS-p"" was developed in 2018. In addition to the elements corresponding to the three conventional domains of physical, cognitive and emotional health constituting the adult PICS, the PICS-p include a domain of ""social health"" of children and their families. This latter aspect is justified by the fact that serious illness affects the social functioning of children and their families; that is, reintegration with friends at school, their social capital and the impact on the work of parents caring for a sick child. These social health problems, intertwined with morbidity in other health domains, can have a further negative impact on the quality of child development and survival. A variety of recovery trajectories for surviving children and their families have been described in the PICS - p framework: improvement, deterioration, vacillation or plateau in the days or decades following PICU discharge. The available data, although still limited, suggest that the situations of children and parents with respect to PICS are more heterogeneous than those of adult post-resuscitation survivors. A 2017 review described the physical, neurocognitive and psychological outcomes in several cohorts of children who survived critical illness in intensive care, with most cohorts investigating a single health domain (physical or neurocognitive or psychological morbidity). In the same review, the authors found that outcomes were more common in younger children, from families with low socioeconomic status, with more invasive procedures or interventions, with high doses of benzodiazepines and narcotics, and varied by disease type.

A wide range of psychological complications have also been described in families. While research on siblings is limited, one review reported prevalence of acute stress, post-traumatic stress symptoms, anxiety and significant depression in parents after their child's discharge from intensive care (between 10 and 84% varying between studies and symptoms). Psychological symptoms persist for several months. Risk factors for long-term problems include unexpected admission to the ICU and the number of medical interventions performed there, limited social support and negative memories of the ICU stay. It should be noted that post-traumatic symptoms in children are associated with parental symptoms.

Today, in the majority of hospitals, there is no specific procedure for the prevention or management of PICS-p. In a recent editorial, pediatricians questioned the role of everyone in promoting a full recovery of children after intensive care: intensive care professionals, families, pediatricians in downstream services, professionals in rehabilitation, psychology or psychiatry, or ambulatory medicine; without giving a single answer.

Our hypothesis is that PICS-p affects a significant proportion of children and families and that identifying its prevalence and associated needs through a descriptive survey will improve management beyond research.

The aim of this study is to describe (in nature and frequency) the alterations in health defined by the WHO of children who have been admitted to PICU and that might constitute a PICS-p.

We will perform a prospective cohort study in Robert-Debré University Hospital including children admitted to the PICU and hospitalized more than 72 hours.

We will include children with an unplanned hospitalization for acute complication of sickle cell disease (such as acute chest syndrome or vaso-occlusive crisis), acute asthma or sepsis for more than 72 hours and aged from 3 to 17 years.

We plan to include 40 patients admitted to the PICU as well as 40 controls admitted to the general pediatrics unit or the pneumology unit without PICU admission, matched on diagnosis, age range and period.

Patients with intellectual retardation or with no health insurance coverage will be excluded.

The primary endpoint will be the prevalence of children that had been admitted to PICU and reporting cognitive, psychological, physical and social impairments measured by questionnaire and medical record data collection on the day before discharge and at the routine post-hospitalization visit.

Secondary objectives will be to study the risk factors for PICS-P, to compare alterations in cognitive, psychological, physical and social domains in children with the same diagnosis and age not admitted to the PICU during their hospitalization.

In order to this, we will measure the association with the PICU stay characteristics, parental experience and social characteristics of families. We will also report the prevalence of children not admitted in PICU and reporting cognitive, psychological, physical and social impairments measured by questionnaire and medical record data collection on the day before discharge and at the routine post-hospitalization visit.

Children will be included on the occasion of an unscheduled hospitalization in general pediatrics or pediatric pulmonology. After informing the family and collecting the consent form, the parents and/or the child will be asked to fill in a questionnaire the day before discharge. Patients and their parents will be given questionnaires the day before discharge and during the first follow-up consultation between 1and 3 months after hospital discharge. In fact, medical consultations are systematically carried out on these children to validate the discharge of patients from hospital (either in the general pediatric department or in the pediatric pneumology department) and a follow-up consultation is systematically carried out between 1 and 3 months after discharge.

Questionnaires will include the Pediatric Symptom Checklist (PSC) long version (Assessment of cognitive, psychological and social domains - 35 items scored from 0 to 2) reported by parents for children under 8 years and by the patients for children older than 8 years. older), the physical items of Pediatric Quality of Life scale (8 items scored from 0 to 4) and a parent self-questionnaire (including relationship to child, annual income, household composition, understanding and use of the French language, highest diploma of mother and father, social support (""How many people can you really count on when you need help?"")) and a parental mental health self-assessment (PHQ-8). The selected questionnaires are validated and available in French and English. One of them will be available in pictorial form (PSC). The most appropriate translation will be offered to the family. If the family has difficulty understanding and/or reading French, it will be systematically proposed to complete the questionnaires with a clinical study technician trained in research who will offer assistance in completing the questionnaires with the ""voice"" function of the Google translate tool, in the family's preferred language. The results of these questionnaires may eventually lead to changes in the patient's usual care, as for ethical reasons, families will be provided with psychological support contacts to contact if they feel the need, and any disorders identified will be managed.

In addition to questionnaires, additional data will be collected in the computerized medical record: child gender, child date of birth, diagnosis, date of diagnosis, number of previous unscheduled hospitalizations, reason for hospitalization, number of previous PICU visits, unpredictability of ICU admission, reason for PICU visit, length of stay in PICU, number and nature of medical interventions performed in PICU (non-invasive ventilation, intubation, mechanical ventilation, central catheter placement, arterial catheter placement, intraosseous catheter placement, pleural puncture, chest tube placement…), sedations used (molecules, number), withdrawal syndrome, delirium, date of discharge from PICU, number and nature of medical interventions performed outside the PICU, date of admission to general pediatrics or pneumology unit and dat of discharge from hospital, mode of discharge (home, transfer to other facilities including rehabilitation centers), psychologic disorders during stay, reported sequelae including respiratory and neurologic ones.

The analyses will be descriptive (description of the nature and frequency of alterations) and comparative (between children who have or have not been in PICU). Univariate tests will be performed to identify possible risk factors for post intensive care syndrome.

Statistics will be carried out on SAS 9.4 software.

ELIGIBILITY:
Inclusion Criteria:

* Children with a diagnosis of an acute complication of sickle cell disease such as acute chest syndrome or vaso-occlusive crisis, asthma attack or sepsis Unscheduled hospitalization at Robert Debré Hospital For more than 72 hours
* Ages 3 to 17

Exclusion Criteria:

* transfers (not possible to collect information the day before discharge)
* Participant unable or unwilling to comply with study procedures (including persons who do not speak French and cannot be assisted by a third party who speaks French)

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children hospitalised (not planned) for asthma, SCD, sepsis in a tertiary pediatric hospital; with or without PICU care
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-10-19 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
prevalence of children reporting Post Intensive Care Syndrome in pediatrics measured by questionnaire and medical record data collection | 4 months
  questionnaire and medical record data collection

CONTACTS AND LOCATIONS:
Overall Officials: Michael LEVY, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Robert Debré Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No